CLINICAL TRIAL: NCT04623294
Title: Online Noninvasive Assessment of Human Brain Death and Deep Coma by Near-infrared Spectroscopy With Protocol at Varied Fraction of Inspired O2
Brief Title: Online Noninvasive Assessment of Human Brain Death and Deep Coma by Near-infrared Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ting Li, Full professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NIRS for brain death and coma
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Brain Death; Coma
Keywords: Brain death; Deep coma; Oxygen metabolism; Near infrared spectroscopy
MeSH Terms: conditions — Brain Death; Coma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Brain death patients for HLH Oxygen: Brain-dead patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of high-low-high procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by the NIRS instrument for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of high-low-high procedure
- Brain death patients for LHL Oxygen: Brain-dead patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of low-high-low procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by the NIRS instrument for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of low-high-low procedure
- Deep coma patients for HLH Oxygen: Deep coma patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of high-low-high procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by the NIRS instrument for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of high-low-high procedure
- Deep coma patients for LHL Oxygen: Deep coma patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of low-high-low procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by the NIRS instrument for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of low-high-low procedure
- Healthy people for HLH Oxygen: Healthy people were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of high-low-high procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of high-low-high procedure
- Healthy people for LHL Oxygen: Healthy people were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of low-high-low procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of low-high-low procedure

INTERVENTIONS:
Procedure: Oxygen supply of high-low-high procedure — The protocol consisted of 1-hour resting, 3-minute baseline measurement, half-hour measurement at 60% FIO2(phase I, high oxygen), half-hour measurement at 40% FIO2 (phase II, low oxygen) and half-hour measurement at 60% FIO2 (phase III, high oxygen).
  Device: Optical monitor for hemodynamic parameter. Near infrared spectroscopy instrument was attached on the subjects' forehead to detect the changes of hemodynamic parameters.
  Groups: Brain death patients for HLH Oxygen; Deep coma patients for HLH Oxygen; Healthy people for HLH Oxygen
Procedure: Oxygen supply of low-high-low procedure — The protocol consisted of 1- hour resting, 3-minute baseline measurement, half-hour measurement at 40% FIO2 (phase I, low oxygen), half-hour measurement at 60% FIO2 (phase II, high oxygen) and half-hour measurement at 40% FIO2 (phase III, low oxygen).
  Device: Optical monitor for hemodynamic parameter. Near infrared spectroscopy instrument was attached on the subjects' forehead to detect the changes of hemodynamic parameters.
  Groups: Brain death patients for LHL Oxygen; Deep coma patients for LHL Oxygen; Healthy people for LHL Oxygen

SUMMARY:
This study aims to assess brain death and deep coma with the self-made near infrared spectroscopy (NIRS) instrument. The investigators used the noninvasive method to monitor the Δ[HbO2] (the concentration changes in oxy-hemoglobin) and Δ[Hb] (the concentration changes in deoxy-hemoglobin) in the region around the forehead of medically evaluated participating patients and healthy subjects. A multiple-phase protocol at varied fraction of inspired O2 were utilized during the assessment.

DETAILED DESCRIPTION:
Brain death is an irreversible loss of all brain functions, while deep coma is a profound state of unconsciousness associated with depressed cerebral activity. Timely distinguishing the two states is crucial for saving patients. The noninvasive, sensitive, universally available, and timely ancillary method to assess brain death and deep coma has not been established. This study aims to explore a noninvasive and straightforward way in brain death and deep coma online assessment. The changes of hemodynamic parameters including oxyhemoglobin (HbO2) and deoxyhemoglobin (Hb) were detected by near infrared spectroscopy instrument attached on the forehead of participators. A multiple-phase protocol at varied fraction of inspired O2(FIO2) were utilized during the assessment. Then the investigators compared the multiple physiological parameters changes among different groups at different FIO2.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had brain death or serious brain trauma.
* Patients who have deep coma with autonomous respiration according to GCS coma Scale
* Healthy people who are interested in optical assessment of hemodynamic parameters

Exclusion Criteria:

* Patients who are in pregnancy or have plan to conception.
* Patients who have vertebra surgery or have plan of surgery.
* Patients who are inappropriate to join this trial judged by the radiologists or specialists.
* AIDS, Active Hepatitis, Tuberculosis, Syphilis
* Patients who regularly take anticoagulants, antiplatelet drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals of any gender. Hired from Intensive Care Center of Sichuan Provincial People's Hospital，Shanghai Xinhua Hospital and Tianjin Huanhu Hospital
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Δ[HbO2] | 1 day during the whole experiment
  The changes of oxyhemoglobin concentrations in prefrontal cortex.
Δ[Hb] | 1 day during the whole experiment
  The changes of deoxyhemoglobin concentrations in prefrontal cortex.

SECONDARY OUTCOMES:
Heart rate | 1 day during the whole experiment
  Heart rate of patient recorded by bed-side physiological monitor.
Blood pressure | 1 day during the whole experiment
  Blood pressure of patient recorded by bed-side physiological monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- NIRS assessment for brain death, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Pan B, Huang C, Fang X, Huang X, Li T. Noninvasive and sensitive optical assessment of brain death. J Biophotonics. 2019 Mar;12(3):e201800240. doi: 10.1002/jbio.201800240. Epub 2018 Dec 13. PMID 30379409